CLINICAL TRIAL: NCT06817538
Title: Investigation of the Effects of Dual Task Training on Dual Task Performance in Individuals With Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gözde Yagci (Gür), Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HUTez_001
Record Dates: First submitted 2024-05-16; First posted 2025-02-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Scoliosis
Keywords: adolescent; dual task; scoliosis; gait parameters
MeSH Terms: conditions — Scoliosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Non-drug clinical research and method comparison clinical research
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Task Group (Other): Control
  Interventions: Behavioral: Physiotherapy/Exercise Program
- Dual Task Group (Other): Study
  Interventions: Behavioral: Physiotherapy/Exercise Program

INTERVENTIONS:
Behavioral: Physiotherapy/Exercise Program — Arm 1: Scoliosis-Specific Exercises Combined with Dual-Task Cognitive Training Participants with idiopathic scoliosis in this group received scoliosis-specific physiotherapeutic exercises combined with dual-task cognitive training. The intervention included motor exercises performed on balance boards and stability trainers to enhance postural control. While engaging in these motor exercises, participants simultaneously performed cognitive tasks such as word recall, identifying cities or countries starting with a given letter, and other memory-based games. This dual-task approach aimed to improve both motor and cognitive functions.
  Arm 2: Scoliosis-Specific and Motor Exercises Only
  Participants with idiopathic scoliosis in this group performed scoliosis-specific physiotherapeutic exercises along with motor exercises aimed at improving postural stability. The motor exercises were conducted using balance boards and stability trainers, focusing solely on physical performance without the

SUMMARY:
In this study, "Single Task" and "Dual Task" groups will be formed in individuals aged 10-18 years with scoliosis. For 12 weeks, scoliosis-specific three-dimensional exercises will be applied to both groups. The Single Task group will receive only motor exercise training, while the Dual Task group will receive both motor and cognitive exercise training. At the end of the study, the dual-task performance of both groups will be evaluated and the effects of dual task training on individuals with scoliosis will be analyzed.

DETAILED DESCRIPTION:
Scoliosis is a term used to describe changes in the shape and position of the spine and chest cage. Essentially, scoliosis involves lateral deviation and rotations of the vertebrae, accompanied by changes in the sagittal plane, creating a three-dimensional deformity. The progressive nature of scoliotic deformity underscores the importance of controlling these components through conservative methods. Without control, scoliosis can lead to postural, balance, and locomotor disorders due to compromised sensory integrity and inadequate proprioceptive feedback. Despite compromised postural control and continuity in individuals with Adolescent Idiopathic Scoliosis (AIS), maintaining daily life activities and body orientation is crucial for controlling the progression of scoliosis. The daily routine of individuals with AIS often involves simultaneous engagement in postural control alongside other daily activities. These routines and exercises frequently incorporate dual-task components. Our study aims to examine the effectiveness of single-task and dual-task walking and balance exercises in individuals with scoliosis, as well as their contributions to scoliosis-specific assessments

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 10-16
2. Individuals with idiopathic scoliosis
3. Individuals with curve degrees between 10 and 40
4. Individuals with a body mass index of less than 30 kg\m2.
5. Be willing to participate in the tests and have the cognitive ability to complete the tests.

Exclusion Criteria:

1. Having other types of scoliosis other than idiopathic scoliosis
2. Individuals with previous scoliosis or any spine-related conservative treatment or surgery
3. Acute (fracture, surgery); cardiovascular system (heart failure, arrhythmia...); nervous system diseases (epilepsy, vertigo...); sensory organs (vision or hearing loss...); musculoskeletal disorders (rheumatism, hypermobility syndrome...)
4. Taking any regular medication that may affect balance (ssri, psycholeptic, anti-epileptic medication...)
5. Playing sports at a professional level
6. Using a brace, starting to use a brace

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Single Motor - Cadence | From baseline assessment to post-intervention at 12 weeks (after 12 exercise sessions, one session per week)
  10 meter walking test. Measurements will begin with the participant's first step from the starting line and will end as they cross the finish line. Each participant will complete three trials, during which the step count and duration will be recorded. Based on these evaluations cadence (steps/min) will be calculated.
Single Motor - Step Lengths | From baseline assessment to post-intervention at 12 weeks (after 12 exercise sessions, one session per week)
  10 meter walking test. Measurements will begin with the participant's first step from the starting line and will end as they cross the finish line. Each participant will complete three trials, during which the step count and duration will be recorded. Based on these evaluations step lengths (m) will be calculated.
Single Motor - Walking Speed | From baseline assessment to post-intervention at 12 weeks (after 12 exercise sessions, one session per week)
  10 meter walking test. Measurements will begin with the participant's first step from the starting line and will end as they cross the finish line. Each participant will complete three trials, during which the step count and duration will be recorded. Based on these evaluations, walking speed (m/min) will be calculated.
Single Cognitive | From baseline assessment to post-intervention at 12 weeks (after 12 exercise sessions, one session per week)
  Stroop Test
Dual-Task ( Number) | From baseline assessment to post-intervention at 12 weeks (after 12 exercise sessions, one session per week).
  Giving specific cognitive tasks during a 10m walk. These cognitive tasks will be counting backwards in 7's from a random number between 50-100.
Dual-Task (Letter) | From baseline assessment to post-intervention at 12 weeks (after 12 exercise sessions, one session per week).
  Participants will read a 5-letter word backward during a 10-meter walk. Each word will be provided randomly, and participants will be instructed to articulate the letters of the word in reverse order while walking.

SECONDARY OUTCOMES:
Body Asymmetry and Posture Assessments | Baseline measurements conducted at the initial assessment. Participants will undergo a 12-week exercise intervention, with one session per week. Post-treatment assessments will be conducted immediately after completing the 12 sessions at the 12th week.
  Anterior and Posterior Trunk Symmetry Index
Scoliosis-specific assessments 2 | Baseline measurements conducted at the initial assessment. Participants will undergo a 12-week exercise intervention, with one session per week. Post-treatment assessments will be conducted immediately after completing the 12 sessions at the 12th week.
  Anterior Trunk Rotation. The ATR is measured with the help of a scoliometer (inclinometer), a scoliosis measuring device, which evaluates the rotation of the trunk in degrees with the patient in a forward-bent position (Adam's Test position)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy and Rehabilitation, Hacettepe, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No